CLINICAL TRIAL: NCT03098979
Title: A Multicenter, Randomized, Placebo-controlled, Parallel Group, Double Blind, Dose-finding Phase II Trial to Study the Efficacy, Safety, Pharmacokinetics and Pharmacodynamic Effects of the Oral Partial Adenosine A1 Receptor Agonist Neladenoson Bialanate Over 20 Weeks in Patients With Chronic Heart Failure and Preserved Ejection Fraction
Brief Title: A Trial to Study Neladenoson Bialanate Over 20 Weeks in Patients With Chronic Heart Failure With Preserved Ejection Fraction
Acronym: PANACHE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17582; 2016-004062-26 (EudraCT Number)
Record Dates: First submitted 2017-03-15; First posted 2017-04-04 (Actual); Results first posted 2019-07-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Heart Failure
Keywords: Chronic Heart Failure; Heart Failure with Preserved Ejection Fraction
MeSH Terms: conditions — Heart Failure | interventions — neladenoson bialanate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Neladenoson bialanate (BAY1067197) (5 mg) (Experimental): Chronic heart failure with preserved ejection fraction
  Interventions: Drug: Neladenoson bialanate (BAY1067197)
- Neladenoson bialanate (BAY1067197) (10 mg) (Experimental): Chronic heart failure with preserved ejection fraction
  Interventions: Drug: Neladenoson bialanate (BAY1067197)
- Neladenoson bialanate (BAY1067197) (20 mg) (Experimental): Chronic heart failure with preserved ejection fraction
  Interventions: Drug: Neladenoson bialanate (BAY1067197)
- Neladenoson bialanate (BAY1067197) (30 mg) (Experimental): Chronic heart failure with preserved ejection fraction
  Interventions: Drug: Neladenoson bialanate (BAY1067197)
- Neladenoson bialanate (BAY1067197) (40 mg) (Experimental): Chronic heart failure with preserved ejection fraction
  Interventions: Drug: Neladenoson bialanate (BAY1067197)
- Placebo (Placebo Comparator): Chronic heart failure with preserved ejection fraction
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Neladenoson bialanate (BAY1067197) — 5 mg orally once daily for 20 weeks
  Arms: Neladenoson bialanate (BAY1067197) (5 mg)
Drug: Neladenoson bialanate (BAY1067197) — 10 mg orally once daily for 20 weeks
  Arms: Neladenoson bialanate (BAY1067197) (10 mg)
Drug: Neladenoson bialanate (BAY1067197) — 20 mg orally once daily for 20 weeks
  Arms: Neladenoson bialanate (BAY1067197) (20 mg)
Drug: Neladenoson bialanate (BAY1067197) — 30 mg orally once daily for 20 weeks
  Arms: Neladenoson bialanate (BAY1067197) (30 mg)
Drug: Neladenoson bialanate (BAY1067197) — 40 mg orally once daily for 20 weeks
  Arms: Neladenoson bialanate (BAY1067197) (40 mg)
Drug: Placebo — Orally once daily for 20 weeks
  Arms: Placebo

SUMMARY:
The objective of the study is to find the optimal dose of once daily oral neladenoson bialanate (BAY1067197) when given in addition to appropriate therapy for specific comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 45 years and older
* Diagnosis of chronic heart failure, NYHA (New York Heart Association) class II-IV, LVEF (left ventricular ejection fraction) ≥ 45% and elevated NT-proBNP

Exclusion Criteria:

* Acute decompensated heart failure within the past 4 weeks
* Inability to exercise
* Previous diagnosis of HFrEF (heart failure with reduced ejection fraction) (LVEF < 40%)

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2018-05-23 (Actual); Study Completion 2018-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (76):
- United States (4):
  - Northwestern University, Chicago, Illinois
  - St. Louis Heart & Vascular, PC, St Louis, Missouri
  - BryanLGH Medical Center East, Lincoln, Nebraska
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
- Austria (6):
  - Universitätsklinikum St. Pölten, Sankt Pölten, Lower Austria
  - Medizinische Universität Graz, Graz, Styria
  - Krankenhaus St. Josef Braunau, Braunau am Inn, Upper Austria
  - Krankenhaus der Elisabethinen Linz GmbH, Linz, Upper Austria
  - Allgemeines Krankenhaus der Stadt Wien, Vienna
  - Krankenhaus Hietzing, Vienna
- Belgium (3):
  - Jessa Ziekenhuis, Hasselt
  - CHR de la Citadelle, Liège
  - AZ Delta, Roeselare
- Bulgaria (6):
  - Spec Hosp for Active Treatm in Cardiology Sv Georgi Pernik, Pernik
  - Specialized Hospital for Actrive Treatm of Card - Pleven, Pleven
  - Medical Center Cardiohelp, Sofia
  - NMTH Tzar Boris III, Sofia
  - UMHAT Tsaritsa Joanna-ISUL EAD Sofia, Sofia
  - MCOMH Preventsia-2000, Stara Zagora
- Germany (4):
  - St. Vincenz und Elisabeth Hospital, Kathol. Klinikum Mainz, Mainz, Rhineland-Palatinate
  - Klinische Forschung Dresden GmbH, Dresden, Saxony
  - HELIOS Klinikum Erfurt GmbH, Erfurt, Thuringia
  - Charité Campus Virchow-Klinikum (CVK), Berlin
- Greece (6):
  - KAT General Hospital of Athens, Kifisia / Athens, Attica
  - G. Gennimatas General State Hospital of Athens, Athens
  - General Hospital of Chalkida, Chalcis
  - Konstantopoulio General Hospital of Nea Ionia - Agia Olga, Nea Ionia / Athens
  - Hippokration General Hospital of Thessaloniki, Thessaloniki
  - Asklipieion General Hospital of Voulas, Voula
- Israel (7):
  - Barzilai Medical Center, Ashkelon
  - Hillel Yaffe Medical Center, Hadera
  - Rambam Health Corporation, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah University Hospital Mount Scopus, Jerusalem
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
  - Assaf Harofeh Medical Center, Zrifin
- Italy (7):
  - AAS 3 Friuli Alto Medio Collin, Udine, Friuli Venezia Giulia
  - A.O.U. Sant'Andrea, Rome, Lazio
  - ASST Papa Giovanni XXIII, Bergamo, Lombardy
  - ASST Spedali Civili di Brescia, Brescia, Lombardy
  - A.O. Ordine Mauriziano, Turin, Piedmont
  - A.O.U. di Sassari, Sassari, Sardinia
  - AUSL Toscana Sud-Est, Arezzo, Tuscany
- Japan (14):
  - Chuno kosei Hospital, Sekimachi, Gifu
  - Hyogo Prefectural Amagasaki General Medical Center, Amagasaki, Hyōgo
  - National Hospital Organization Kanazawa Medical Center, Kanazawa, Ishikawa-ken
  - Shonan Fujisawa Tokushukai Hospital, Fujisawa, Kanagawa
  - R.I.A.C Naha City Hospital, Naha, Okinawa
  - Kishiwada Tokushukai Hospital, Kishiwada, Osaka
  - Takatsuki Red Cross Hospital, Takatsuki, Osaka
  - Osaka Medical College Hospital, Takatsuki, Osaka
  - Minamino Cardiovascular Hospital, Hachiōji, Tokyo
  - Tokyo Women's Medical University Hospital, Shinjuku-ku, Tokyo
  - Fukui Prefectural Hospital, Fukui
  - Okayama Rosai Hospital, Okayama
  - Osaka General Medical Center, Osaka
  - Tokushima Prefectural Central Hospital, Tokushima
- Poland (7):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok
  - Szpital Zachodni w Grodzisku Mazowieckim, Grodzisk Mazowiecki
  - Szpital Specjalistyczny im. J. Dietla, Krakow
  - Wojewodzki Specjalistyczny Szpital im. dr Wl. Bieganskiego, Lodz
  - 109 Szpital Wojskowy z przychodnia SPZOZ, Szczecin
  - Szpital Wolski im. dr Anny Gostynskiej SPZOZ, Warsaw
  - IV Wojskowy Szpital Kliniczny z Poliklinika, SPZOZ, Wroclaw
- Portugal (4):
  - CHUC - Hospitais da Universidade de Coimbra, Coimbra
  - CHLO - Hospital São Francisco Xavier, Lisbon
  - Hospital da Luz, Lisbon
  - CHUP, EPE - Hospital de Santo Antonio, Porto
- Spain (8):
  - Hospital Sanitas La Zarzuela, Aravaca, Madrid
  - Hospital Universitario "Virgen de la Arrixaca", El Palmar, Murcia
  - Hospital del Mar, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Clínico Universitario San Carlos, Madrid
  - Hospital Virgen de la Victoria, Málaga
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitari i Politècnic La Fe, Valencia

REFERENCES:
- [Derived] Shah SJ, Voors AA, McMurray JJV, Kitzman DW, Viethen T, Bomfim Wirtz A, Huang E, Pap AF, Solomon SD. Effect of Neladenoson Bialanate on Exercise Capacity Among Patients With Heart Failure With Preserved Ejection Fraction: A Randomized Clinical Trial. JAMA. 2019 Jun 4;321(21):2101-2112. doi: 10.1001/jama.2019.6717. PMID 31162568

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 76 study centers in 12 countries, between 10 May 2017 (first patient first visit) and 20 June 2018 (last patient last visit)
Pre-assignment Details: A total of 339 subjects entered the screening period, of whom 34 withdrew before randomization. The remaining 305 subjects were randomized and received at least one dose of study drug
Groups:
- Placebo: Subjects received placebo matched to neladenoson bialanate tablets orally for 20 weeks
- Neladenoson Bialanate 5 mg: Subjects received 5 milligrams (mg) of neladenoson bialanate tablets orally for 20 weeks
- Neladenoson Bialanate 10 mg: Subjects received 10 mg of neladenoson bialanate tablets orally for 20 weeks
- Neladenoson Bialanate 20 mg: Subjects received 20 mg of neladenoson bialanate tablets orally for 20 weeks
- Neladenoson Bialanate 30 mg: Subjects received 30 mg of neladenoson bialanate tablets orally for 20 weeks
- Neladenoson Bialanate 40 mg: Subjects received 40 mg of neladenoson bialanate tablets orally for 20 weeks
Period: Overall Study
Arm/Group | Placebo | Neladenoson Bialanate 5 mg | Neladenoson Bialanate 10 mg | Neladenoson Bialanate 20 mg | Neladenoson Bialanate 30 mg | Neladenoson Bialanate 40 mg
Started | 76 | 27 | 50 | 51 | 50 | 51
Completed | 70 | 25 | 46 | 46 | 41 | 47
Not Completed | 6 | 2 | 4 | 5 | 9 | 4
Not completed — Adverse Event | 1 | 0 | 1 | 4 | 6 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 1 | 1 | 2 | 1
Not completed — Death | 1 | 0 | 2 | 0 | 1 | 0
Not completed — Physician Decision | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Non-compliance | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Neladenoson Bialanate 5 mg | Neladenoson Bialanate 10 mg | Neladenoson Bialanate 20 mg | Neladenoson Bialanate 30 mg | Neladenoson Bialanate 40 mg | Total
Number analyzed (Participants) | 76 | 27 | 50 | 51 | 50 | 51 | 305
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.1 (8.0) | 74.3 (9.3) | 73.5 (9.9) | 71.4 (6.8) | 76 (9.4) | 73.7 (8.3) | 73.6 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 16 | 26 | 21 | 32 | 29 | 160
  Male | 40 | 11 | 24 | 30 | 18 | 22 | 145
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 0 | 0 | 0 | 0 | 2
  Not Hispanic or Latino | 73 | 27 | 49 | 51 | 50 | 50 | 300
  Unknown or Not Reported | 1 | 0 | 1 | 0 | 0 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 9 | 3 | 6 | 5 | 5 | 5 | 33
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 0 | 0 | 1 | 0 | 1 | 5
  White | 64 | 24 | 44 | 45 | 45 | 45 | 267
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
LVEF [Mean (Standard Deviation); unit: percentage of blood ejected] — Left ventricular ejection fraction (LVEF) is defined as the fraction of blood being pumped out of the left ventricle of the heart with each contraction. Population: Included subjects with valid baseline value for this characteristic
  percentage of blood ejected
    number analyzed (Participants) | 45 | 20 | 32 | 32 | 32 | 33 | 194
    (all) | 57.09 (8.68) | 56.54 (9.62) | 53.78 (11.6) | 57.3 (10.4) | 59.43 (8.72) | 52.3 (12.76) | 56.09 (10.5)
NT-proBNP [Median (Full Range); unit: pg/ml] — N-terminal pro-hormone b-type natriuretic peptide Population: Included subjects with valid baseline value for this characteristic
  pg/ml
    number analyzed (Participants) | 63 | 23 | 44 | 42 | 39 | 44 | 255
    (all) | 882.0 [54 to 3034] | 1013.0 [136 to 5709] | 1000.0 [116 to 3547] | 834.5 [173 to 6003] | 626.0 [78 to 3043] | 886.5 [60 to 8170] | 869.0 [54 to 8170]
NYHA class [Count of Participants; unit: Participants] — NYHA classes: I: No limitation of physical activity (PA). Ordinary PA does not cause undue fatigue, palpitation, dyspnea, or anginal pain II: Slight limitation of PA; comfortable at rest. Ordinary PA results in fatigue, palpitation, dyspnea, or anginal pain III: Marked limitation of PA; comfortable at rest. Less than ordinary PA causes fatigue, palpitation, dyspnea, or anginal pain IV: Inability to carry on any PA without discomfort. Symptoms of heart failure or the anginal syndrome may be present even at rest. If any PA is undertaken, discomfort is increased
  Participants
    II | 61 | 23 | 37 | 41 | 31 | 39 | 232
    III/IV | 15 | 4 | 13 | 10 | 19 | 12 | 73
Medical history: diabetes [Count of Participants; unit: Participants] — Subjects with medical history of Type 2 diabetes mellitus
  Participants | 36 | 7 | 23 | 20 | 22 | 21 | 129
Medical history: Atrial fibrillation [Count of Participants; unit: Participants] — Subjects with medical history of Atrial fibrillation
  Participants | 28 | 10 | 18 | 19 | 20 | 21 | 116
Medical history: hypertension [Count of Participants; unit: Participants] — Subjects with medical history of hypertension
  Participants | 66 | 25 | 45 | 45 | 46 | 42 | 269
eGFR [Mean (Standard Deviation); unit: mL/min/1.73 square meter] — eGFR = estimated glomerular filtration rate
  mL/min/1.73 square meter | 62.0 (17.9) | 52.6 (17.1) | 61.0 (24.2) | 57.1 (17.3) | 57.5 (18.2) | 60.0 (17.5) | 59.1 (18.9)
6MWD [Mean (Standard Deviation); unit: meter] — 6MWD = six-minute walking distance
  meter | 322.8 (97.1) | 311.6 (108.2) | 295.8 (110.4) | 324.5 (105) | 321.1 (93.4) | 347.2 (94.5) | 321.5 (101)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in 6-minute Walking Distance (6MWD) After 20 Weeks of Treatment
Description: The 6MWD test is designed to evaluate a subject's exercise capacity while performing an everyday activity.
Time Frame: Baseline, and up to 20 weeks of treatment
Population: Per-protocol set (PPS): Included all full analysis set (FAS) population subjects without validity findings for this outcome measure, and it also included subjects who were censored due to cardiovascular (CV) death or hospitalization for heart failure (HF) that prevented assessment of efficacy at 20 weeks.
Measure: Mean (Standard Deviation); unit: meter
Arm/Group | Placebo | Neladenoson Bialanate 5 mg | Neladenoson Bialanate 10 mg | Neladenoson Bialanate 20 mg | Neladenoson Bialanate 30 mg | Neladenoson Bialanate 40 mg
Number analyzed (Participants) | 65 | 22 | 44 | 41 | 34 | 37
meter
  Value at baseline | 329 (95) | 306 (117) | 300 (109) | 328 (105) | 321 (101) | 363 (83)
  Change from baseline to Week 20 | 1.89 (49.5) | 24.8 (72.4) | 27.2 (90.0) | 14.6 (54.1) | 16.3 (55.4) | 10.7 (60.2)
Statistical Analysis 1: Comparison: Placebo vs Neladenoson Bialanate 5 mg vs Neladenoson Bialanate 10 mg vs Neladenoson Bialanate 20 mg vs Neladenoson Bialanate 30 mg vs Neladenoson Bialanate 40 mg; Test type: Superiority; p = 0.5183, MCP-Mod method — Linear dose-response shape: The multiple comparison procedures (MCP) approach was applied to calculate the adjusted one-sided p-values of the contrast test; Dose response relationship was assessed using the MCP-Mod method combining MCP principles with modeling techniques
Statistical Analysis 2: Comparison: Placebo vs Neladenoson Bialanate 5 mg vs Neladenoson Bialanate 10 mg vs Neladenoson Bialanate 20 mg vs Neladenoson Bialanate 30 mg vs Neladenoson Bialanate 40 mg; Test type: Superiority; p = 0.3300, MCP-Mod method — Sigmoidal Emax 1 dose-response shape: The MCP approach was applied to calculate the adjusted one-sided p-values of the contrast test; Dose response relationship was assessed using the MCP-Mod method combining MCP principles with modeling techniques
Statistical Analysis 3: Comparison: Placebo vs Neladenoson Bialanate 5 mg vs Neladenoson Bialanate 10 mg vs Neladenoson Bialanate 20 mg vs Neladenoson Bialanate 30 mg vs Neladenoson Bialanate 40 mg; Test type: Superiority; p = 0.6232, MCP-Mod method — Sigmoidal Emax 2 dose-response shape: The MCP approach was applied to calculate the adjusted one-sided p-values of the contrast test; Dose response relationship was assessed using the MCP-Mod method combining MCP principles with modeling techniques
Statistical Analysis 4: Comparison: Placebo vs Neladenoson Bialanate 5 mg vs Neladenoson Bialanate 10 mg vs Neladenoson Bialanate 20 mg vs Neladenoson Bialanate 30 mg vs Neladenoson Bialanate 40 mg; Test type: Superiority; p = 0.0918, MCP-Mod method — Emax dose-response shape: The MCP approach was applied to calculate the adjusted one-sided p-values of the contrast test; Dose response relationship was assessed using the MCP-Mod method combining MCP principles with modeling techniques
Statistical Analysis 5: Comparison: Placebo vs Neladenoson Bialanate 5 mg vs Neladenoson Bialanate 10 mg vs Neladenoson Bialanate 20 mg vs Neladenoson Bialanate 30 mg vs Neladenoson Bialanate 40 mg; Test type: Superiority; p = 0.2701, MCP-Mod method — Quadratic dose-response shape: The MCP approach was applied to calculate the adjusted one-sided p-values of the contrast test; Dose response relationship was assessed using the MCP-Mod method combining MCP principles with modeling techniques

2. Secondary Outcome: Change From Baseline in Average Weekly Percentage of Maximum Possible Recorded Activity Intensity
Description: AVIVO™ Mobile Patient Management System, a wearable wireless device worn by the subject, was used to monitor subjects' cardiovascular status. The patient's everyday physical activity e.g. duration, intensity, was also tracked by the AVIVO device. For Activity Intensity, the Unit of Measure is "percentage of maximum activity", and length of intervals is "daily".
Time Frame: Baseline, and up to 20 weeks of treatment
Population: Per-protocol set (PPS): Included all full analysis set (FAS) population subjects without validity findings for this outcome measure
Measure: Mean (Standard Deviation); unit: percentage of maximum activity
Arm/Group | Placebo | Neladenoson Bialanate 5 mg | Neladenoson Bialanate 10 mg | Neladenoson Bialanate 20 mg | Neladenoson Bialanate 30 mg | Neladenoson Bialanate 40 mg
Number analyzed (Participants) | 56 | 20 | 39 | 35 | 32 | 33
percentage of maximum activity
  Value at visit Baseline | 2.83 (1.03) | 2.76 (0.72) | 2.83 (0.95) | 2.51 (0.91) | 2.61 (0.94) | 2.43 (0.57)
  Change from baseline at Week 20: number analyzed (Participants) | 52 | 20 | 34 | 33 | 30 | 32
  Change from baseline at Week 20 | -0.19 (0.58) | -0.25 (0.51) | -0.12 (0.58) | -0.08 (0.67) | -0.18 (0.57) | -0.14 (0.57)

3. Secondary Outcome: Measured Values (Log Transformed) and Absolute Change in NT-proBNP From Baseline to 20 Weeks
Description: NT-proBNP = N-terminal pro-hormone b-type natriuretic peptide
Time Frame: Baseline, and up to 20 weeks of treatment
Population: as for outcome 2
Measure: Median (Full Range); unit: log (pg/ml)
Arm/Group | Placebo | Neladenoson Bialanate 5 mg | Neladenoson Bialanate 10 mg | Neladenoson Bialanate 20 mg | Neladenoson Bialanate 30 mg | Neladenoson Bialanate 40 mg
Number analyzed (Participants) | 62 | 21 | 44 | 39 | 33 | 36
log (pg/ml)
  Value at baseline | 6.80 [4.0 to 8.0] | 6.78 [4.9 to 8.1] | 6.81 [4.8 to 8.2] | 6.73 [5.2 to 8.7] | 6.68 [4.5 to 8.0] | 6.64 [4.1 to 8.8]
  Absolute change from baseline to Week 20: number analyzed (Participants) | 60 | 20 | 43 | 38 | 32 | 36
  Absolute change from baseline to Week 20 | -0.07 [-1.3 to 1.6] | 0.08 [-3.0 to 0.9] | 0.13 [-1.7 to 1.6] | 0.06 [-1.2 to 2.3] | 0.09 [-1.3 to 0.9] | 0.19 [-1.0 to 2.9]

4. Secondary Outcome: Measured Values (Log-transformed) and Absolute Change in High Sensitivity Troponin T (Hs-TNT) From Baseline to 20 Weeks
Description: High sensitivity troponin T (hs-TNT) was measured
Time Frame: Baseline, and up to 20 weeks of treatment
Population: as for outcome 2
Measure: Median (Full Range); unit: log(pg/mL)
Arm/Group | Placebo | Neladenoson Bialanate 5 mg | Neladenoson Bialanate 10 mg | Neladenoson Bialanate 20 mg | Neladenoson Bialanate 30 mg | Neladenoson Bialanate 40 mg
Number analyzed (Participants) | 63 | 22 | 44 | 38 | 33 | 37
log(pg/mL)
  Value at baseline | 2.92 [1.9 to 4.4] | 3.25 [1.9 to 4.7] | 2.95 [1.9 to 4.7] | 2.76 [1.9 to 4.2] | 2.73 [1.9 to 3.9] | 2.76 [1.9 to 4.8]
  Absolute change from baseline to Week 20: number analyzed (Participants) | 60 | 22 | 44 | 38 | 33 | 36
  Absolute change from baseline to Week 20 | 0.00 [-1.4 to 1.6] | 0.02 [-0.9 to 0.9] | 0.00 [-0.7 to 1.1] | 0.12 [-0.8 to 1.5] | 0.13 [-0.4 to 1.2] | 0.01 [-0.8 to 0.9]

5. Secondary Outcome: Measured Values and Absolute Change in 3 Scores From Kansas City Cardiomyopathy Questionnaire (KCCQ) From Baseline to 20 Weeks: Overall Summary Score, Physical Limitation Score and Total Symptom Score
Description: The KCCQ is the leading health-related quality-of-life measure for patients with chronic heart failure (CHF). It is a 23-item questionnaire that independently measures the impact of patient's heart failure (HF), or its treatment, on 7 distinct domains: 1) Symptom Frequency 2) Symptom Burden 3) Physical Limitation 4) Quality of Life 5) Social Limitations 6) Self-efficacy 7) Symptoms Stability.
  Overall summary score= mean score of (symptom frequency + symptom burden+ physical limitation + quality of life + social limitation); scores on a scale of 0 to 100, higher scores means better outcome; Physical Limitation: scores on a scale of 0 to 100, higher scores means better outcome; Total symptom score=mean score of (symptom frequency + symptom burden): scores on a scale of 0 to 100, higher scores means better outcome.
  Positive change means improvement and negative change means deterioration.
Time Frame: Baseline, and up to 20 weeks of treatment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Neladenoson Bialanate 5 mg | Neladenoson Bialanate 10 mg | Neladenoson Bialanate 20 mg | Neladenoson Bialanate 30 mg | Neladenoson Bialanate 40 mg
Number analyzed (Participants) | 65 | 22 | 44 | 41 | 34 | 37
scores on a scale
  Overall Summary Score Baseline | 69.19 (18.02) | 64.75 (23.99) | 66.42 (21.21) | 64.57 (20.73) | 63.67 (17.76) | 64.65 (18.07)
  Overall Summary Score Change from baseline: number analyzed (Participants) | 65 | 22 | 44 | 41 | 33 | 37
  Overall Summary Score Change from baseline | 3.38 (13.55) | 7.04 (17.24) | -1.33 (20.61) | 3.73 (13.03) | 0.27 (14.83) | 2.25 (14.25)
  Physical Limitation Score Baseline | 69.07 (19.43) | 63.18 (25.24) | 68.03 (22.79) | 69.35 (22.64) | 64.53 (22.47) | 63.12 (23.44)
  Physical Limitation Score Change from baseline: number analyzed (Participants) | 65 | 22 | 43 | 40 | 33 | 37
  Physical Limitation Score Change from baseline | 2.18 (17.54) | 1.40 (17.62) | -1.34 (22.56) | 0.92 (14.65) | -3.75 (22.10) | 2.17 (17.32)
  Total Symptom Score Baseline | 76.78 (19.64) | 72.25 (21.73) | 68.99 (23.13) | 69.99 (20.18) | 68.00 (20.09) | 71.03 (18.80)
  Total Symptom Score Change from baseline: number analyzed (Participants) | 65 | 22 | 44 | 41 | 33 | 37
  Total Symptom Score Change from baseline | 2.96 (15.85) | 5.82 (17.51) | 0.14 (19.08) | 3.56 (14.04) | 2.54 (16.79) | 2.62 (16.04)

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to 26 weeks
Groups:
- Neladenoson Bialanate 5mg: Subjects received 5 mg of neladenoson bialanate tablets orally for 20 weeks.
- Neladenoson Bialanate 10mg: Subjects received 10 mg of neladenoson bialanate tablets orally for 20 weeks.
- Neladenoson Bialanate 20mg: Subjects received 20 mg of neladenoson bialanate tablets orally for 20 weeks.
- Neladenoson Bialanate 30mg: Subjects received 30 mg of neladenoson bialanate tablets orally for 20 weeks.
- Neladenoson Bialanate 40mg: Subjects received 40 mg of neladenoson bialanate tablets orally for 20 weeks.
Arm/Group | Placebo | Neladenoson Bialanate 5mg | Neladenoson Bialanate 10mg | Neladenoson Bialanate 20mg | Neladenoson Bialanate 30mg | Neladenoson Bialanate 40mg
All-Cause Mortality (participants affected / at risk) | 2/76 | 0/27 | 2/50 | 1/51 | 1/50 | 1/51
Serious Adverse Events (participants affected / at risk) | 21/76 | 9/27 | 11/50 | 11/51 | 14/50 | 16/51
Other Adverse Events (participants affected / at risk) | 24/76 | 13/27 | 14/50 | 22/51 | 17/50 | 24/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=76) | Neladenoson Bialanate 5mg (N=27) | Neladenoson Bialanate 10mg (N=50) | Neladenoson Bialanate 20mg (N=51) | Neladenoson Bialanate 30mg (N=50) | Neladenoson Bialanate 40mg (N=51)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 2 (2) | 2 (2) | 3 (3) | 4 (4) | 2 (2) | 7 (8)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 3 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinoatrial block (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis media chronic (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arteriogram coronary (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza A virus test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intraventricular haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Basal ganglia haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insertion of ambulatory peritoneal catheter (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hysterosalpingectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device dislocation (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=76) | Neladenoson Bialanate 5mg (N=27) | Neladenoson Bialanate 10mg (N=50) | Neladenoson Bialanate 20mg (N=51) | Neladenoson Bialanate 30mg (N=50) | Neladenoson Bialanate 40mg (N=51)
Atrial fibrillation (Cardiac disorders) | 5 (5) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 4 (6)
Cardiac failure (Cardiac disorders) | 5 (5) | 2 (3) | 3 (3) | 6 (9) | 1 (1) | 3 (3)
Ventricular tachycardia (Cardiac disorders) | 3 (5) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 5 (6) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 2 (2)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (4) | 0 (0)
Nasopharyngitis (Infections and infestations) | 5 (6) | 1 (1) | 3 (3) | 3 (3) | 2 (3) | 4 (5)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 1 (2) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 3 (4) | 3 (4)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (5) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 4 (4) | 2 (3) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 5 (5)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 2 (2) | 5 (6) | 3 (3) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 1 (1) | 0 (0) | 4 (6) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Material for public dissemination will be submitted to the Sponsor for review at least thirty (30) days prior to submission for publication, public dissemination, or review by a publication committee. If Sponsor does not respond within this period Institution and/or the Principal Investigator is/are free to proceed with the intended publication or presentation without further delay

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-06-15): https://cdn.clinicaltrials.gov/large-docs/79/NCT03098979/SAP_000.pdf
  • Study Protocol (2017-02-14): https://cdn.clinicaltrials.gov/large-docs/79/NCT03098979/Prot_001.pdf